CLINICAL TRIAL: NCT02450994
Title: Dexamethasone for Prophylaxis of Sleep Related Breathing Disturbances in Patients With Chronic Obstructive Pulmonary Disease (COPD) Travelling to Altitude
Brief Title: Effect of Dexamethasone on Sleep Related Breathing Disturbances in Patients With COPD at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EK15-2015_V1
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; lung; treatment; sleep
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 4 mg capsules, twice per day, orally
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo capsules twice per day, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Dexamethasone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of dexamethasone in preventing sleep related breathing disturbances in lowlanders with chronic obstructive lung disease travelling from 700 m to 3200 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of dexamethasone prophylaxis in sleep related breathing disturbances in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (700m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Dexamethasone 2x4mg/day (or placebo), will be administered before departure at 700 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease (COPD), GOLD grade 1-2
* Living at low altitude (<800m)

Exclusion Criteria:

* COPD exacerbation
* severe COPD, GOLD grade 3 or 4
* arterial oxygen saturation <92% at low altitude (<800 m)
* Diabetes, uncontrolled cardiovascular disease such as systemic arterial hypertension, coronary artery disease; previous stroke; pneumothorax in the last 2 months, untreated or symptomatic peptic ulcer disease, glaucoma, obstructive sleep apnea.
* Internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day).
* pregnant or nursing patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | night 1 at 3200 m
  Difference in mean nocturnal oxygen saturation between dexamethasone and placebo group

SECONDARY OUTCOMES:
Oxygen desaturation index | night 1 at 3200 m
  Difference in oxygen desaturation index (>3%) between dexamethasone and placebo group
Mean nocturnal oxygen saturation measured by pulse oximetry | night 2 at 3200 m
  Difference in mean nocturnal oxygen saturation between dexamethasone and placebo group
Apnea/hypopnea index | night 2 at 3200 m
  Difference in mean apneas/hypopneas per hour between the dexamethasone and placebo group
Apnea/hypopnea index | night 1 at 3200 m
  Difference in mean apneas/hypopneas per hour between the dexamethasone and placebo group
Oxygen desaturation index | night 2 at 3200 m
  Difference in oxygen desaturation index (>3%) between dexamethasone and placebo group
Mean nocturnal oxygen saturation measured by pulse oximetry | night 1 at 700 m
  Difference in mean nocturnal oxygen saturation between dexamethasone and placebo group
Oxygen desaturation index | night 1 at 700 m
  Difference in oxygen desaturation index (>3%) between dexamethasone and placebo group
Apnea/hypopnea index | night 1 at 700 m
  Difference in mean apneas/hypopneas per hour between the dexamethasone and placebo group
Psychomotor vigilance test reaction time | day 2 at 700 m
  Difference in reaction time during psychomotor vigilance test between dexamethasone and placebo group
Subjective sleepiness | day 2 at 700 m
  Difference in subjective sleepiness and sleep quality assessed by a visual analog scale between dexamethasone and placebo group
Subjective sleepiness | day 2 at 3200 m
  Difference in subjective sleepiness and sleep quality assessed by a visual analog scale between dexamethasone and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Furian M, Lichtblau M, Aeschbacher SS, Estebesova B, Emilov B, Sheraliev U, Marazhapov NH, Mademilov M, Osmonov B, Bisang M, Ulrich S, Latshang TD, Ulrich S, Sooronbaev TM, Bloch KE. Effect of Dexamethasone on Nocturnal Oxygenation in Lowlanders With Chronic Obstructive Pulmonary Disease Traveling to 3100 Meters: A Randomized Clinical Trial. JAMA Netw Open. 2019 Feb 1;2(2):e190067. doi: 10.1001/jamanetworkopen.2019.0067. PMID 30794302